CLINICAL TRIAL: NCT00390858
Title: A 4-year Extension to a Phase II a Multicenter Study Evaluating Long-term Safety, Tolerability, Pharmacokinetics and Effects on Liver Iron Concentration of Repeated Doses of 10 mg/kg/Day of Deferasirox in Pediatric Patients With Transfusion Dependent β-thalassemia Major.
Brief Title: A 4-year Extension Study to Core 1-year Study of Iron Chelation Therapy With Deferasirox in β-thalassemia Major Pediatric Patients With Transfusional Iron Overload.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0106E1
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Transfusional Iron Overload; β-thalassemia Major; Pediatric Rare Anemia
Keywords: β-thalassemia major; iron overload; deferasirox; pediatric rare anemia
MeSH Terms: conditions — Iron Overload | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental): Initial dose of 10 mg/kg, dose modifications of ± 5 or 10 mg/kg were based on participant response.
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — Deferasirox in children from 1 to 18 years old was given orally once daily, 30 minutes prior to breakfast. An initial daily dose of 10 mg/kg was used during the 1-year core study. In this 4-year extension study dose modifications of ± 5 or 10 mg/kg were based on safety parameters and on increasing or decreasing Liver Iron Concentration (LIC), and serum ferritin. Deferasirox was available as 125 mg, 250 mg and 500 mg tablets.
  Other Names: ICL670

SUMMARY:
In this 4-year extension study the safety, efficacy and and pharmacokinetics of deferasirox in regularly transfused pediatric patients with β-thalassemia major was assessed. Patients who successfully completed the main 1 year trial (NCT00390858) were eligible to continue in this extension trial and receive chelation therapy with deferasirox for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the planned 12-month core trial, (NCT00390858).
* Female patients who have reached menarche and who were sexually active were to use double-barrier contraception, oral contraceptive plus barrier contraceptive, or must have undergone clinically documented total hysterectomy and/or ovariectomy, or tubal ligation.
* Written informed consent obtained from the patient, and/or from the parent or legal guardian in accordance with the national legislation.

Exclusion Criteria:

* Pregnant or breast feeding patients
* Patients with a history of non-compliance to medical regimens and patients who are considered by the investigator as potentially unreliable.

Other protocol-defined exclusion criteria may apply.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2003-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gianluca Forni, Study Director — Novartis Pharmaceuticals; Prof. Renzo Galanello, Study Director — Novartis Pharmaceuticals; Prof. Antonio Piga, Study Director — Novartis Pharmaceuticals; Dr. Yves Bertrand, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Lyon, France
- Italy (3):
  - Novartis Investigative Site, Cagliari
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Torino

RESULTS

PARTICIPANT FLOW:
Groups:
- Children ( < 12 Years); Adolescents ( ≧12 Years): Deferasirox was given orally once daily, 30 minutes prior to breakfast. An initial daily dose of 10 mg/kg was used during the 1-year core study. In this 4-year extension study dose modifications of ± 5 or 10 mg/kg were based on safety parameters (e.g. renal and hematology) and whether Liver Iron Concentration (LIC), and serum ferritin were increasing or decreasing
Period: Overall Study
Arm/Group | Children ( < 12 Years) | Adolescents ( ≧12 Years)
Started | 20 (20 participants started the Core Study) | 20 (20 Participants started the Core Study)
Completed Core & Entered Extension Study | 19 | 20
Completed | 11 (11 participants Completed the Extension Study) | 13 (13 Participants completed the Extension Study)
Not Completed | 9 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Children (<12 Years); Adolescents ( ≧12 Years): Deferasirox was given orally once daily, 30 minutes prior to breakfast. An initial daily dose of 10 mg/kg was used during the 1-year core study. In this 4-year extension study dose modifications of ± 5 or 10 mg/kg were based on safety parameters (e.g. renal and hematology) and whether Liver Iron Concentration (LIC), and serum ferritin were increasing or decreasing
- Total: Total of all reporting groups
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.7 (2.83) | 14.1 (1.64) | 10.4 (4.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events by Primary System Organ Class (SOC)
Description: Safety parameters were measured by the number and type of adverse events (AEs). An adverse event is any untoward medical occurence in a patient administered a medicinal product that does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign ( for example, an abnormal laboratory finding), symptom or disease temporally associated with the use of the medicinal product, whether or not this is associated with the use of this medicinal product.
Time Frame: 4 year extension + core 1 year
Population: The safety set comprising of all the 40 patients who received at least one dose of deferasirox during the core or extension study was used in all analyses.
Measure: Number; unit: participants
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years)
Number analyzed (Participants) | 20 | 20
participants
  Patients with at least one Adverse Event (AE) | 20 | 20
  General disorders & administration site conditions | 19 | 20
  Respiratory, thoracic & mediastinal disorders | 19 | 17
  Gastrointestinal disorders | 18 | 17
  Infections & infestations | 18 | 17
  Musculoskeletal & connective tissue disorders | 12 | 15
  Investigations | 13 | 10
  Nervous system disorders | 9 | 13
  Skin & subcutaneous tissue disorders | 12 | 8
  Injury, poisoning & procedural complications | 11 | 8
  Ear & labyrinth disorders | 9 | 8
  Metabolism & nutrition disorders | 6 | 10
  Eye disorders | 6 | 9
  Renal & urinary disorders | 3 | 6
  Hepatobiliary disorders | 1 | 7
  Reproductive system & breast disorders | 0 | 8
  Cardiac disorders | 1 | 5
  Blood & lymphatic system disorders | 1 | 5
  Psychiatric disorders | 2 | 4
  Immune system disorders | 0 | 2
  Surgical & medical procedures | 0 | 3
  Endocrine disorders | 1 | 1
  Vascular disorders | 0 | 2
  Congenital, familial & genetic disorders | 1 | 0

2. Primary Outcome: Change in Liver Iron Concentration (LIC)
Description: Change in Liver Iron Concentration [LIC] measured by means of SQUID (Superconducting Quantum Interference Device). LIC is expressed in milligrams of iron per gram of liver dry weight (mg Fe/g dw)
Time Frame: Baseline of Core Study to End of Extension Study, up to 5 years.
Population: The safety set was used for all analyses. This comprised of all 40 patients who received at least one dose of deferasirox during the core or extension study.
Measure: Mean (Standard Deviation); unit: mg Fe/g dw
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years)
Number analyzed (Participants) | 20 | 20
mg Fe/g dw
  Core Baseline LIC (n = 20, 20) | 6.25 (2.507) | 5.73 (2.185)
  End of Extension LIC (n=19, 20) | 5.46 (3.192) | 4.66 (3.533)
  Change from Baseline LIC (n=19, 20) | -0.9 (3.85) | -1.10 (3.03)

3. Secondary Outcome: Total Body Iron Elimination (TBIE) Rate (mg/kg/Day)
Description: Total Iron Body Elimination (TBIE) Rate [mg/kg/Day] was calculated for each patient based on SQUID ( Superconducting Quantum Interference Device) results.
Time Frame: Baseline of Core Study to End of Extension Study, up to 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/kg/Day
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years)
Number analyzed (Participants) | 20 | 20
mg/kg/Day
  Core Baseline TBIE (n=19, 20) | 0.4292 (0.06454) | 0.4083 (0.07158)
  End of Extension TBIE (n=11,14) | 0.4939 (0.05175) | 0.4286 (0.06370)

4. Secondary Outcome: Relative Change in Serum Ferritin Level
Description: Serum levels were drawn at the baseline of the Core Study up to 18 months of the Extension Study. Levels were analyzed for serum ferritin measured in micrograms per Liter. Relative change (%) in serum ferritin level was assessed from Baseline to Extension 18 months. Relative Change = 1 - (Change in ferritin level from Baseline/Baseline level) x 100.
Time Frame: Baseline of Core Study to Extension 18 months, up to 2.5 years.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years)
Number analyzed (Participants) | 20 | 20
percent change | 62.4 (53.47) | 54.9 (64.64)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Core Study Baseline to Extension End of Study, up to 5 years.
Groups:
- Children (<12 Years); Adolescents ( ≧12 Years): Deferasirox was given orally once daily, 30 minutes prior to breakfast. An initial daily dose of 10 mg/kg was used during the 1-year core study. In this 4-year extension study dose modifications of ± 5 or 10 mg/kg were based on safety parameters ( renal and hematology) and whether Liver Iron Concentration (LIC) and serum ferritin were increasing or decreasing
Arm/Group | Children (<12 Years) | Adolescents ( ≧12 Years)
Serious Adverse Events (participants affected / at risk) | 4/20 | 8/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children (<12 Years) (N=20) | Adolescents ( ≧12 Years) (N=20)
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 2
Splenectomy (Surgical and medical procedures) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Children (<12 Years) (N=20) | Adolescents ( ≧12 Years) (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 4
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Talipes (Congenital, familial and genetic disorders) | 1 | 0
Auricular pseudocyst (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 8 | 4
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3
Growth hormone deficiency (Endocrine disorders) | 1 | 0
Hypogonadism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 3 | 4
Conjunctivitis allergic (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Hypermetropia (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Ocular icterus (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 15 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 8
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Dental caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 3 | 4
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 2
Intestinal congestion (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 10
Odynophagia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 12 | 9
Asthenia (General disorders) | 7 | 8
Chest pain (General disorders) | 1 | 3
Cyst (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 3
Influenza like illness (General disorders) | 3 | 1
Pyrexia (General disorders) | 18 | 16
Suprapubic pain (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 4
Jaundice (Hepatobiliary disorders) | 0 | 1
Allergy to plants (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 5 | 5
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 9 | 2
Fungal infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 10 | 8
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital infection female (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 7 | 11
Laryngitis (Infections and infestations) | 2 | 1
Leptospirosis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 2
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 2 | 2
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 12 | 10
Pharyngotonsillitis (Infections and infestations) | 1 | 4
Pyoderma (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 17 | 13
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tinea versicolour (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 3 | 5
Tooth abscess (Infections and infestations) | 2 | 1
Tracheitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Varicella (Infections and infestations) | 5 | 1
Vulvitis (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 3 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 1
Vertebral injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Beta 2 microglobulin urine increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2
Blood folate decreased (Investigations) | 1 | 0
Blood homocysteine increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Glomerular filtration rate abnormal (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Protein C decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 8 | 2
Urinary casts (Investigations) | 1 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 1
Vitamin E decreased (Investigations) | 2 | 4
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperinsulinism (Metabolism and nutrition disorders) | 0 | 1
Hypozincaemia (Metabolism and nutrition disorders) | 1 | 1
Vitamin C deficiency (Metabolism and nutrition disorders) | 1 | 2
Zinc deficiency (Metabolism and nutrition disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 3
Aphonia (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 12
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Nervousness (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal colic (Renal and urinary disorders) | 0 | 2
Amenorrhoea (Reproductive system and breast disorders) | 0 | 3
Breast discomfort (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 4
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.